CLINICAL TRIAL: NCT00977132
Title: Phase II Study for the Determination of Efficacy and Tolerability of the Combination of Valproic Acid and Lenalidomide in the Treatment of Patients With Myelodysplastic Syndrome With Favorable Risk Profile
Brief Title: Efficacy and Tolerability of the Combination of Valproic Acid and Lenalidomide in the Treatment of Patients With Myelodysplastic Syndrome
Acronym: VALENA
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: delayed recruitment
Sponsor: Heinrich-Heine University, Duesseldorf (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Valena-Study
Record Dates: First submitted 2009-09-14; First posted 2009-09-15 (Estimated); Last update posted 2015-03-18 (Estimated); Status verified 2015-03

CONDITIONS: Myelodysplastic Syndrome MDS
Keywords: Myelodysplastic Syndromes; Valproic acid; Lenalidomide
MeSH Terms: conditions — Anemia, Refractory, with Excess of Blasts; Myelodysplastic Syndromes | interventions — Lenalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Lenalidomide (Experimental): Lenalidomid in combination valproic acid
  Interventions: Drug: Valproic aicd; Drug: Lenalidomide

INTERVENTIONS:
Drug: Valproic aicd — Treatment with VPA starts at day1, the dose ist slowly increase according to the following scheme
  day morning dose midday dose evening dose contents of 1 tablet
  1+2 0 0 1 500 mg
  3+4 ½ 0 1 500 mg
  5+6 1 0 1 500 mg
  7+8 1 ½ 1 500 mg
  9+10 1 1 1 500 mg
  11+12 1 1 1 500 mg
  In the morning of day 13 trough level of VPA will be checked. The target range will be 50-110 µg/l. The dose of VPA will be adjusted depending on the trough level. In the first eight weeks of therapy weekly controls of VPA levels are required. Thereafter, VPA levels will be checked every four weeks.
Drug: Lenalidomide — 5 mg/day, continuous therapy
  Dosing will be in the morning at approximately the same time each day. Capsules may be taken before or after a meal.
  Only one cycle of study drug (28 days) will be supplied to the patient every four weeks
  Other Names: Revlimid

SUMMARY:
As part of a palliative therapy concept, feasibility, toxicity, and effectiveness of treatment with the combination of Valproic acid and lenalidomide in Myelodysplastic Syndrome patients with a favorable risk profile will be investigated.

DETAILED DESCRIPTION:
Treatment will be administered as continuous therapy, i.e. it should be taken on each day as described below without treatment interruption as long as no criteria for termination of treatment are met. After two years the primary endpoint will be evaluated. Non-responders will be taken off study after 4 months of therapy. Patients who relapse after an initial response to study treatment can receive one attempt to re-start therapy after a short duration of discontinuation.

Treatment with Valproic Acid starts at day 1. The dose of Valproic Acid is slowly increased. In the morning of day 13 trough level of Valproic Acid will be checked. The target range will be 50-110 µg/l. The dose of Valproic Acid will be adjusted depending on the trough level.

In the first eight weeks of therapy weekly controls of Valproic Acid levels are required. Thereafter, Valproic Acid levels will be checked every four weeks.

The planned dose of lenalidomide is 10 mg/day, orally as continuous therapy. Dosing will be in the morning at approximately the same time each day. Capsules may be taken before or after a meal. In the course of the study the dose will be adjusted to the results of the blood count.

Only one cycle of study drug (28 days) will be supplied to the patient every four weeks.

Patients experiencing adverse events may need study treatment modifications.

During treatment with study medication weekly control visits for the detection of adverse events are required during the first eight weeks, thereafter the patient must be seen every four weeks.

Therapeutic success is evaluated in 4-weekly intervals. Bone marrow will be examined after 12 weeks and after 48 weeks or in case of premature study termination

ELIGIBILITY:
Inclusion Criteria:

* Cytologically/histologically confirmed primary myelodysplastic syndrome (pMDS) with a favorable risk profile, i.e., low or intermediate I risk group according to IPSS (<10% blasts, no unfavorable karyotype)
* platelet count ≥50.000/µl
* absolute neutrophil count ≥1.000/µl
* age ≥18 years at the time of signing the informed consent form
* Karnofsky performance status > 50%
* written informed consent to participate
* erythropoietin level > 200 mU/ml or failure of previous therapy with erythropoietin
* patients in whom allogeneic bone marrow transplantation, treatment with growth factors or immune therapy is not possible due to medical or biologic reasons or patients in whom such a therapy would be possible but who do not agree to such a therapy for personal reasons
* females of childbearing potential (FCBP, see page 23) must agree to one reliable form of contraception or to practice complete abstinence from heterosexual intercourse during the following time periods related to this study: 1) for at least 4 weeks before starting study drug; 2) while participating in the study, even during treatment interruptions; and 3) for at least 4 weeks after discontinuation from the study.

Exclusion Criteria:

* patients with 5q deletion
* MDS treated with experimental therapy or chemotherapy within 4 weeks prior to start of treatment with study drugs
* previous treatment of MDS with valproic acid or lenalidomide as monotherapy patients suitable for chemotherapy, therapy with growth factors or allogeneic bone marrow transplantation and who are willing to start such a therapy
* hypersensitivity to thalidomide
* insufficient liver function (bilirubin, AST or ALT > 2 x ULN)
* hepatic disease [details see full protocol]
* markedly impaired renal function (serum creatinine > 2mg/dl)
* pregnancy, breast feeding, lactation, refusal to use safe contraceptive methods during the study
* psychiatric disease or addiction with impaired ability to act and make decisions according to one's free will
* participation in another interventional study 4 weeks prior to or during this study
* known hypersensitivity or allergies to one of the study drugs or their ingredients
* plasmatic coagulation disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2009-10; Primary Completion 2013-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
hematologic success | 5 years

SECONDARY OUTCOMES:
toxicity and safety | 5 years
Progression free survival | 5 years
overall survival | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Norbert Gattermann, Professor, Study Director — Department of Hematology, Oncology and Clinical Immunology
Locations (6):
- Germany (6):
  - Medizinische Universitätsklinik Freiburg, Abteilung Innere Medizini, Freiburg im Breisgau, Baden Würtemberg
  - Universitätsklinikum Ulm, Klinik für Innere Medizin III, Ulm, Bavaria
  - Georg-August-Universität,Universitätsklinikum - Abteilung Hämatologie und Onkologie, Göttingen, Lower Saxony
  - St. Johannes Hospital Duisburg, Duisburg, North Rhine-Westphalia
  - Heinrich-Heine-University Duesseldorf, Department of Hematology, Oncology and Clinical Immunology, Düsseldorf, North Rhine-Westphalia
  - Universitätsklinikum Carl Gustav Carus an der TU Dresden, Medizinische Klinik und Poliklinik I, Dresden, Saxony